CLINICAL TRIAL: NCT04293120
Title: Training Anticipatory Postural Adjustments Among People With Neurodevelopmental Disabilities
Brief Title: Training Balance Among People With Neurodevelopmental Disabilities
Acronym: TAPAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID restrictions prevented recruitmetn
Sponsor: University of Hartford (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Mary Gannotti, Professor, University of Hartford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO19020012
Record Dates: First submitted 2020-02-10; First posted 2020-03-03 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Posture; Balance; Cerebral Palsy; Autism; Down Syndrome
MeSH Terms: conditions — Cerebral Palsy; Autistic Disorder; Down Syndrome

STUDY DESIGN:
Intervention Model Description: Case control, matched on gender, age, and BMI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental): Training 4 sessions over a one week time period of 180 catches/stops with a medicine ball.
  Interventions: Other: Training with weighted ball

INTERVENTIONS:
Other: Training with weighted ball — Participants will stop or catch a weighted ball

SUMMARY:
This study is a case control pilot study to investigate the impact of a short-term intervention on training anticipatory postural adjustments in a population of people with neurodevelopmental disabilities.

DETAILED DESCRIPTION:
Data will be collected by using a weighted pendulum to provide a posterior perturbation to test subjects' postural reactions pre and post-intervention. Intervention will include four sessions of weighted ball tosses/weighted tether ball stops to improve muscle activation patterns and efficiency. EMG sensors, 3D motion analysis, and force plates will be used to collect the necessary data.

ELIGIBILITY:
Inclusion Criteria:

Participants

1. Able to stand without assistance
2. Diagnosis of cerebral palsy, Down Syndrome, or Autism Spectrum Disorder
3. Able to stop weighted ball without falling
4. Able to follow directions

Controls

1. Able to stand without assistance
2. No neurodeveloopmental disability
3. Able to stop weighted ball without falling
4. Able to follow directions

Exclusion Criteria:

1. Pregnancy
2. Unable to maintain standing when stopping a ball on a rope

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Muscle activation timing | Pre-intervention muscle activation timing will be assessed on the initial visit. Post-intervention muscle activation timing will be assessed immediately after the fourth training session, at most, 7 days later.
  Evaluation in change in muscle activation timing of anterior tibialis, soleus, gastroc, rectus femoris, biceps femoris, rectus abdominis using electromyography

SECONDARY OUTCOMES:
Muscle amplitude response | Pre-intervention muscle amplitude response will be assessed on the initial visit. Post-intervention muscle amplitude response will be assessed immediately after the fourth training session, at most, 7 days later.
  Evaluation in change in amplitude of anterior tibialis, soleus, gastroc, rectus femoris, biceps femoris, rectus abdominis using electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Gannotti, PT, PhD, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No